CLINICAL TRIAL: NCT00799422
Title: Evaluation of Lens Fit, Lens Parameters, and Circumlimbal Conjunctival Staining (CSS) in Normal Patients
Brief Title: Evaluation of Contact Lenses and Conjunctival Staining in Normal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: M-08-02
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Conjunctival Staining
Keywords: Conjunctival Staining; lens parameters; lens fit
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReNu MultiPlus (Active Comparator): ReNu MultiPlus used as specified in the protocol for contact lens care. In this crossover study, ReNu MultiPlus was dispensed in randomized order with Complete Easy Rub and Clear Care. Each product was used for one week with a fresh pair of Acuvue Oasys contact lenses. A 36-hour washout preceded each usage period.
  Interventions: Device: ReNu MultiPlus; Device: Contact lenses
- Complete Easy Rub (Active Comparator): Complete Easy Rub used as specified in the protocol for contact lens care. In this crossover study, Complete Easy Rub was dispensed in randomized order with ReNu MultiPlus and Clear Care. Each product was used for one week with a fresh pair of Acuvue Oasys contact lenses. A 36-hour washout preceded each usage period.
  Interventions: Device: Complete Easy Rub; Device: Contact lenses
- Clear Care (Active Comparator): Clear Care used as specified in the protocol for contact lens care. In this crossover study, Clear Care was dispensed in randomized order with Complete Easy Rub and ReNu MultiPlus. Each product was used for one week with a fresh pair of Acuvue Oasys contact lenses. A 36-hour washout preceded each usage period.
  Interventions: Device: Clear Care; Device: Contact lenses

INTERVENTIONS:
Device: Complete Easy Rub — Commercially marketed contact lens solution for contact lens care
  Other Names: Complete® Easy Rub®
  Arms: Complete Easy Rub
Device: ReNu MultiPlus — Commercially marketed contact lens solution for contact lens care
  Other Names: ReNu MultiPlus®
  Arms: ReNu MultiPlus
Device: Clear Care — Commercially marketed contact lens solution for contact lens care
  Other Names: Clear Care®
  Arms: Clear Care
Device: Contact lenses — Acuvue Oasys silicone hydrogel contact lenses per participant's habitual prescription worn 8-10 hours per day for one week.
  Other Names: ACUVUE® OASYS®

SUMMARY:
The purpose of this study was to investigate contact lens fit, lens parameters, and conjunctival staining in a sample of subjects with various contact lens/solution combinations.

ELIGIBILITY:
Inclusion Criteria:

* Successfully wearing hydrogel and/or silicone hydrogel contact lenses;
* Read, sign, and date informed consent/HIPAA document;
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with habitual spectacles;
* Willing and able to discontinue contact lens wear when requested during the study;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Evidence or history of ocular disease or pathology;
* One functional eye or a monofit lens;
* Use of concomitant topical ocular prescription or over-the-counter ocular medications;
* History of seasonal allergies with significant ocular side effects which may have an adverse impact on contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ramsey, O.D., Study Director — Alcon Research
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this 3-treatment, 3-period, 6-sequence crossover study, each subject received all 3 products in randomized order and used 1 product at a time for a duration of 1 week before switching to the next assigned product. A 36-hour washout preceded each usage period.
Groups:
- ReNu / Complete / Clear Care: ReNu Multiplus, then Complete Easy Rub, then Clear Care, 1 week each
- Complete / Clear Care / ReNu: Complete Easy Rub, then Clear Care, then ReNu MultiPlus, 1 week each
- Clear Care / ReNu / Complete: Clear Care, then ReNu MultiPlus, then Complete Easy Rub, 1 week each
- ReNu / Clear Care / Complete: ReNu MultiPlus, then Clear Care, then Complete Easy Rub, 1 week each
- Complete / ReNu / Clear Care: Complete Easy Rub, then ReNu MultiPlus), then Clear Care, 1 week each
- Clear Care / Complete / ReNu: Clear Care, then Complete Easy Rub, then ReNu MultiPlus, 1 week each
Period: First Week of Wear
Arm/Group | ReNu / Complete / Clear Care | Complete / Clear Care / ReNu | Clear Care / ReNu / Complete | ReNu / Clear Care / Complete | Complete / ReNu / Clear Care | Clear Care / Complete / ReNu
Started | 4 | 4 | 4 | 5 | 4 | 5
Completed | 4 | 4 | 3 | 4 | 4 | 5
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Second Week of Wear
Arm/Group | ReNu / Complete / Clear Care | Complete / Clear Care / ReNu | Clear Care / ReNu / Complete | ReNu / Clear Care / Complete | Complete / ReNu / Clear Care | Clear Care / Complete / ReNu
Started | 4 | 4 | 3 | 3 (One subject discontinued between First and Second 3 weeks (adverse event)) | 4 | 4 (One subject discontinued between First and Second 3 weeks (adverse event))
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Week of Wear
Arm/Group | ReNu / Complete / Clear Care | Complete / Clear Care / ReNu | Clear Care / ReNu / Complete | ReNu / Clear Care / Complete | Complete / ReNu / Clear Care | Clear Care / Complete / ReNu
Started | 4 | 4 | 3 | 3 | 4 | 4
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Baseline characteristics are presented for all participants completing all three treatment sequences.
Arm/Group | Overall
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Circumlimbal Conjunctival Staining Score
Description: Circumlimbal conjunctival staining was expressed as the sum of the individual scores observed across all of the evaluated regions of the eye. The bulbar conjunctiva was assessed by the investigator utilizing a slit-lamp and lissamine green ophthalmic dye. Staining coverage was scored separately in each of four regions (nasal, temporal, inferior, and superior) using a 4-point clinical grading scale (grade 0-3), where Grade 0 = No staining present; Grade 1 = Slight staining present; Grade 2 = Moderate staining present; and Grade 3 = Dense staining present. The scores for the four regions were summed, with a sum score range of 0-12. A lower score represents a more desirable outcome.
Time Frame: 1 week
Population: This reporting group includes all participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- ReNu MultiPlus: ReNu MultiPlus used for one week as specified in the protocol with study contact lenses.
- Complete Easy Rub: Complete Easy Rub used for one week as specified in the protocol with study contact lenses.
- Clear Care: Clear Care used for one week as specified in the protocol with study contact lenses.
Arm/Group | ReNu MultiPlus | Complete Easy Rub | Clear Care
Number analyzed (Participants) | 22 | 22 | 22
Units on a scale | 6.39 (2.30) | 5.55 (2.94) | 5.68 (1.91)

2. Secondary Outcome: Mean Change From Dispense (Day 0) in Lens Base Curve at 1 Week
Description: Lens base curve at dispense was as listed on product label: 8.4 millimeters (mm). Lens base curve at 1 week was as measured after lens removal. A negative number represented a steepening of the base curve.
Time Frame: Dispense (Day 0), 1 week
Population: This reporting group includes all participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ReNu MultiPlus | Complete Easy Rub | Clear Care
Number analyzed (Participants) | 22 | 22 | 22
mm | -0.25 (0.16) | -0.27 (0.17) | -0.25 (0.15)

3. Secondary Outcome: Mean Change From Dispense (Day 0) in Lens Diameter at 1 Week
Description: Lens diameter at dispense was as listed on product label: 14.0 mm. Lens diameter at 1 week was as measured after lens removal. A positive number indicated a widening of lens diameter.
Time Frame: Dispense (Day 0), 1 week
Population: This reporting group includes all participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ReNu MultiPlus | Complete Easy Rub | Clear Care
Number analyzed (Participants) | 22 | 22 | 22
mm | 0.15 (0.10) | 0.13 (0.11) | 0.14 (0.10)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | ReNu MultiPlus | Complete Easy Rub | Clear Care
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReNu MultiPlus (N=22) | Complete Easy Rub (N=22) | Clear Care (N=22)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Unrelated to study procedures or study products

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes